CLINICAL TRIAL: NCT05965206
Title: Implementation of a Pharmacist-Based, Post-Chemotherapy Follow-up Clinic
Status: Completed | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Suwicha Limvorasak, PharmD, Cedars-Sinai Medical Center
Other Study IDs: Study00002683
Record Dates: First submitted 2023-07-20; First posted 2023-07-28 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Cancer
Keywords: Pharmacist; Follow up clinic
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention group: Participants receive a follow-up phone call from a pharmacist approximately 7 business days after receiving intravenous chemotherapy infusion
  Interventions: Behavioral: Follow-up phone interview
- Control group: Participants do not receive a follow-up phone call from a pharmacist after receiving intravenous chemotherapy infusion

INTERVENTIONS:
Behavioral: Follow-up phone interview — Follow-up phone interview within 7 business days after receiving intravenous chemotherapy
  Other Names: Follow-up call
  Groups: Intervention group

SUMMARY:
The purpose of this study is to determine the impact of pharmacists on reducing chemotherapy-related side effects by providing education before and after patients receive intravenous chemotherapy at one of Cedars-Sinai outpatient infusion centers.

Participants will be interviewed via telephone within 7 business days after receiving intravenous chemotherapy from the outpatient cancer center infusion clinic.

DETAILED DESCRIPTION:
The study involves participation at a single timepoint only.

Participants who consented to participate and are considered eligible will be interviewed by a pharmacist via phone at approximately 7 business days after receiving intravenous chemotherapy infusion. Phone call will be made between the hours of 9am - 6pm on Monday - Saturday. Calls are anticipated to last between 15 to 20 minutes. Participants will be asked if they have experienced any adverse events since the infusion, whether or not they have had any barriers taking supportive care medications, and if the patient understands how to manage potential adverse events. If applicable, participants will be provided further education on optimizing adverse events, guided on proper medication administration times, and will be provided with non-pharmacological clinical pearls to minimize chemotherapy-related side effects and optimize supportive care management.

If unable to reach the participant or caregiver after three attempts, the participant will be considered ineligible. Participants can decline participation at any time during the phone call.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Diagnosed with cancer and is receiving treatment with intravenous chemotherapy
* Treatment initiated at Cedars-Sinai Cancer Samuel Oschin Cancer Center (SOCC) or Cedars-Sinai Cancer Beverly Hills (CSCBH)
* English-speaking or lives with English-speaking person
* Access to a working phone

Exclusion Criteria:

* Received follow-up calls through other specialty pharmacy program
* History of infusion related reactions
* Declined participation on follow-up interview
* Age less than 18 years old
* Non-English speaking
* Electronic health record flagged for research opt out

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult cancer patients who initiated treatment with intravenous chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-07-20 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Hospital admission related to chemotherapy within 30-day post treatment | 30 days after receiving the first intravenous chemotherapy
  Number of hospital admission related to chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Suwicha Limvorasak, PharmD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patel SD, Nguyen PAA, Bachler M, Atkinson B. Implementation of postdischarge follow-up telephone calls at a comprehensive cancer center. Am J Health Syst Pharm. 2017 Jun 1;74(11 Supplement 2):S42-S46. doi: 10.2146/ajhp160805. PMID 28506976
- [Background] Nguyen PAA, Enwere E, Gautreaux S, Lin H, Tverdek F, Lu M, Cao H, Chase J, Roux R. Impact of a pharmacy-driven transitions-of-care program on postdischarge healthcare utilization at a national comprehensive cancer center. Am J Health Syst Pharm. 2018 Sep 15;75(18):1386-1393. doi: 10.2146/ajhp170747. Epub 2018 Jul 31. PMID 30065061
- [Result] Cebollero J, LaFollette JA, Walton SM, Adams Curry M. Evaluation of a Pharmacist-Developed, Nurse-Driven Protocol for Management of Parenteral Anticancer Therapy Infusion Reactions in an Ambulatory Infusion Center. J Oncol Pharm Pract. 2023 Jun;29(4):802-809. doi: 10.1177/10781552221079855. Epub 2022 Feb 14. PMID 35164607
- [Result] Crannage AJ, Hennessey EK, Challen LM, Stevens AM, Berry TM. Implementation of a Discharge Education Program to Improve Transitions of Care for Patients at High Risk of Medication Errors. Ann Pharmacother. 2020 Jun;54(6):561-566. doi: 10.1177/1060028019896377. Epub 2019 Dec 21. PMID 31868004